CLINICAL TRIAL: NCT02766790
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Study of TA-65MD in Healthy Volunteers Evaluating Immunosenescence and Telomere Length Over a Nine Month Period
Brief Title: Effect of TA-65MD on Healthy Volunteers
Acronym: TA-65MD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Telomerase Activation Sciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 53816
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo taken once daily in the morning and once daily in the evening
  Interventions: Other: Placebo
- TA-65MD 100 units Dose (Active Comparator): TA-65MD 100 units capsule and placebo capsule; one of them will be taken in the a.m. and one of them will be taken in the p.m.
  Interventions: Dietary Supplement: TA-65MD
- TA-65MD 250 units Dose (Active Comparator): TA-65MD 250 units capsule and placebo capsule; one of them will be taken in the a.m. and one of them will be taken in the p.m.
  Interventions: Dietary Supplement: TA-65MD
- TA-65MD 500 units Dose (Active Comparator): TA-65MD 500 units capsule and placebo capsule; one of them will be taken in the a.m. and one of them will be taken in the p.m.
  Interventions: Dietary Supplement: TA-65MD
- TA-65MD 250 units a.m. and p.m. Dose (Active Comparator): Two TA-65MD 250 units capsules; one of them will be taken in the a.m. and one of them will be taken in the p.m.
  Interventions: Dietary Supplement: TA-65MD

INTERVENTIONS:
Dietary Supplement: TA-65MD — TA-65, a purified small molecule extracted from Astragalus root
  Arms: TA-65MD 100 units Dose; TA-65MD 250 units Dose; TA-65MD 250 units a.m. and p.m. Dose; TA-65MD 500 units Dose
Other: Placebo — Placebo, an inactive formulation
  Arms: Placebo

SUMMARY:
TA-65 MD® is pure, natural, plant-based compound that can help maintain or rebuild telomeres. A telomere is a region of repetitive DNA at the end of a chromosome, which protects the end of the chromosome from deterioration. They shorten during cell division and eventually signal an irreversible state of growth arrest known as cellular senescence. The length of a person's telomeres is an indicator of his or her overall health status; short telomeres have been associated with cellular aging and dysfunction.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the effects of TA-65 MD® on telomere length and on immunosenescence in subjects who have had 9 months of twice daily TA-65 MD® administration, compared to placebo. TA Sciences has developed different doses of TA-65® . The study intends to determine effect of four different doses of TA-65 MD® in terms of biomarkers, telomere length and overall health and sleep status.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males or females, based on medical history and current status.
2. Ages 45-75 years of age (inclusive at the time of Screening).
3. Voluntary consent and methods completion of a signed ICF (informed consent form).
4. BMI that is 18 to 40 kg/m2 (inclusive at the time of Screening).
5. Subjects who are able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions.

   -

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. History of HIV, Hepatitis B, or Hepatitis C.
3. Females who are pregnant, planning to become pregnant during the study, or breastfeeding.
4. Recent or current medical condition that might significantly affect a pharmacodynamic response or compromise the safety of the subject or impact the validity of the study results in the opinion of the Investigator. (e.g., conditions that require taking diuretic medications and/or cardiac stimulants.)
5. Intake of the investigational product within 30 days prior to screening visit.
6. History of an allergic reaction to the study products or ingredient(s) or to comparable products in the opinion of the Investigator.
7. History of drug or alcohol addiction or abuse within 1 year prior to Day -1 product administration through end of study (EOS).
8. Donation of blood within 30 days or plasma within 7 days, prior to Day -1 product administration through EOS.
9. Intolerance to venipuncture or an inability to swallow capsules.

   -

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percent of Immunesenescent cells | 9 months
  Percent of CD3+/CD8+/CD28-, CD3+/CD8+/CD95-, CD8+/CD28-, CD8+/CD95- from whole blood will be measured at baseline and at 9 months. Change in the percent levels of immunesenescent cells in each group compared to baseline and placebo will be evaluated.

SECONDARY OUTCOMES:
clinical laboratory markers | 9 months
  Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Serum creatinine will be measured at screening and at the end of the study. Standard reference range will be followed for these markers.
Telomere length | 9 months
  The change in telomere length in kilobase pair (kb) in each group will be evaluated from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Burkindine, D.O, Principal Investigator — QPS Holdings LLC
Locations (1):
- QPS Bio-Kinetic, LLC, Springfeild, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided